CLINICAL TRIAL: NCT01510288
Title: A Phase 1 Dose Escalation Trial of Ipilimumab in Combination With CG1940 and CG8711 in Patients With Metastatic Hormone-Refractory Prostate Cancer
Brief Title: Phase 1 Trial of Ipilimumab and GVAX in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated because Cell Genesys stopped all activities for GVAX.
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Cell Genesys (Industry); Medarex (Industry)
Responsible Party: Principal Investigator, A.J.M. van den Eertwegh, Dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-0016
Record Dates: First submitted 2012-01-04; First posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Prostate Cancer
Keywords: GVAX; Ipilimumab; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab and GVAX (Experimental)
  Interventions: Drug: GVAX and ipilimumab

INTERVENTIONS:
Drug: GVAX and ipilimumab — All patients receive a 500 million cell priming dose of granulocyte-macrophage colony-stimulating factor-transduced allogeneic prostate cancer cells (GVAX) intradermally on day 1 followed by bi-weekly intradermal injections of 300 million cells for a 24 week period. The vaccinations are combined with monthly intravenous administrations of ipilimumab. The dose-escalation part of this study will be performed using the standard 3+3 phase-I trial design. Patients will be enrolled in cohorts of three; each cohort will receive an escalating dose of ipilimumab at 0•3, 1•0, 3•0 or 5•0 mg/kg. Sixteen patients will be treated in an expansion cohort with GVAX and 3•0 mg/kg ipilimumab.

SUMMARY:
Ipilimumab, an antibody that blocks cytotoxic T-lymphocyte antigen 4, and GVAX have demonstrated anti-tumor activity in prostate cancer. Pre-clinical studies with this combination have demonstrated potent synergy. The purpose of this study is to investigate, using a phase-I 3+3 dose escalation design followed by an expansion cohort, the safety and efficacy of combined treatment with GVAX and ipilimumab in castration-resistant metastatic prostate cancer (CRPC) patients.

DETAILED DESCRIPTION:
A promising immunotherapeutic approach in prostate cancer is whole-cell vaccination. Irradiated allogeneic tumor cells expressing GM-CSF generate a long-lasting and specific anti-tumor immunity in preclinical models. Results from several phase I and II trials showed Prostate GVAX (GVAX) to be well tolerated and suggested improved survival. Cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) is a crucial immune checkpoint molecule that down-regulates T-cell activation and proliferation. Ipilimumab, a fully human monoclonal antibody (IgG1) that blocks CTLA-4, promotes antitumor immunity, and has been demonstrated in two phase III trials to improve overall survival in metastatic melanoma patients. Pre-clinical studies of the anti-CTLA-4 antibody in combination with GM-CSF secreting tumor cell vaccines demonstrated a potent synergy. In this phase I study the investigators examine in CRPC patients whether ipilimumab can be safely combined with GVAX. In addition, the investigators will treat an additional 16 patients at a dose level of 3•0 mg/kg to determine the safety profile and antitumor effects of GVAX and ipilimumab in patients with CRPC.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18-80 years
* Histologic diagnosis of adenocarcinoma of the prostate
* Metastatic prostate cancer deemed to be unresponsive or refractory to hormone therapy
* Detectable metastases by bone scan, CT scan or MRI
* Two consecutive rising PSA values obtained at least two weeks apart and both obtained at least 4-6 weeks after discontinuation of hormone therapy. Second PSA value must be > 5.0 ng/mL. LHRH agonist should not be discontinued.
* Testosterone < 50 ng/dL. Must have had orchiectomy or is currently receiving an LHRH agonist.
* WBC > 3.0 x 109/L, ANC > 1.5 x 109/L, hemoglobin > 6.2 mmol/L, and platelets > 100 x 109/L
* Serum creatinine < 177 umol/L Bilirubin < 1.5 times the upper limit of normal AST < 3 times the upper limit of normal
* ECOG performance status 0-2
* Life expectancy of at least 6 months
* If sexually active, willing to use barrier contraception during the treatment phase of the protocol
* The ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Transitional cell, small cell, neuroendocrine, or squamous cell prostate cancer
* Bone pain severe enough to require routine narcotic analgesia use
* Clinical evidence of brain metastases or history of brain metastases
* Seropositive for HIV, Hepatitis B antigen positive and/or Hepatitis C viremic
* Prior chemotherapy or immunotherapy for prostate cancer
* Radiation therapy within 4 weeks of the first treatment
* Surgery within 4 weeks of the first treatment. Must have recovered from all side effects.
* Flutamide within 4 weeks of the first treatment Megesterol acetate (Megace), finasteride (Proscar), bicalutamide (Casodex),nilutamide, aminoglutethimide, ketoconazole or diethylstilbestrol within 6 weeks of the first treatment.
* Systemic corticosteroid use within 4 weeks of the first treatment
* History of autoimmune disease
* History of another malignancy, except for the following: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, adequately treated Stage I or II cancer currently in complete remission or any other cancer that has been in complete remission for at least 5 years

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-11; Primary Completion 2007-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 7 months

SECONDARY OUTCOMES:
number of patients that have a tumor/PSA response | 7 months
number of patients that will develop a tumor-specific (e.g. PSMA, NY-ESO) antibody response as measured by ELISA | 7 months
the number of patients that have activated T cells and dendritic cells as measured by FACS | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Winald Gerritsen, Prof. MD PhD, Principal Investigator — Amsterdam UMC, location VUmc; Fons van den Eertwegh, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU university medical center, Amsterdam, Netherlands

REFERENCES:
- [Derived] van den Eertwegh AJ, Versluis J, van den Berg HP, Santegoets SJ, van Moorselaar RJ, van der Sluis TM, Gall HE, Harding TC, Jooss K, Lowy I, Pinedo HM, Scheper RJ, Stam AG, von Blomberg BM, de Gruijl TD, Hege K, Sacks N, Gerritsen WR. Combined immunotherapy with granulocyte-macrophage colony-stimulating factor-transduced allogeneic prostate cancer cells and ipilimumab in patients with metastatic castration-resistant prostate cancer: a phase 1 dose-escalation trial. Lancet Oncol. 2012 May;13(5):509-17. doi: 10.1016/S1470-2045(12)70007-4. Epub 2012 Feb 10. PMID 22326922